CLINICAL TRIAL: NCT01990807
Title: Philadelphia -Negative High-risk Children Acute Lymphoblastic Leukemia(ALL) Treatment:Induction Therapy:Vincristine(V),Idarubicin(I),L-asparaginase(L),Dexamethasone(D);Consolidation:V+Daunorubicin(D)+L+D, Methotrexate,Cytarabine
Brief Title: Treatment Protocol of Children With Philadelphia Chromosome Negative High Risk Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Xiaofan Zhu, chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCALL2012
Record Dates: First submitted 2013-11-16; First posted 2013-11-21 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Childhood Acute Lymphoblastic Leukemia; Philadelphia Chromosome, Ph^1^, Absent; B-cell Childhood Acute Lymphoblastic Leukemia
Keywords: high risk; Philadelphia Chromosome absent; Childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Philadelphia Chromosome | interventions — Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Idarubicin(IDA) (Active Comparator): philadelphia negative high -risk ALL : Induction therapy: IDA(6mg/m2/time) one time for each week,altogether 3 times
  Interventions: Drug: Idarubicin(IDA)

INTERVENTIONS:
Drug: Idarubicin(IDA) — 6mg/M2 IV(in the vein) on day 16,22,29 of induction therapy, until progression or unacceptable toxicity develops.
  Other Names: darubicin, IDA, Demethoxydaunor Ubicin

SUMMARY:
The cure rate for childhood acute lymphoblastic leukemia (ALL) has increased significantly in recent decades and expected cure rates now exceed 85%. In recent years, Tyrosine Kinase Inhibitor(TKI) has improved outcome of Philadelphia chromosome positive (Ph+)ALL . But in some high risk groups, The prognosis of patients is still very bad and the relapse rate is high. Clearly, new therapies are urgently needed to prevent and /or treat relapsed ALL.

DETAILED DESCRIPTION:
1. The prognosis of childhood acute lymphoblastic leukemia(ALL) has been increased.
2. Tyrosine Kinase Inhibitor(TKI) has improved Philadelphia chromosome positive (Ph+)ALL treatment outcome.
3. The prognosis of high-risk childhood ALL except for Philadelphia chromosome positive (Ph+)ALL is very bad.

ELIGIBILITY:
Inclusion Criteria:

Children with high-risk ALL Children lower than 18years old

Exclusion Criteria:

Bcr/Abl(+) Children with middle-risk or standard-risk ALL

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
The event free survival of high risk ALL | 2 years

SECONDARY OUTCOMES:
The relapsed rate, death, overall survival | 2 years

OTHER OUTCOMES:
infection rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofan Zhu, MD, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Department of Pediatrics, Institute of Hematology and Blood Disease Hospital, Chinese Academy of Medical Scienses, Tianjin, Tianjin Municipality, China